CLINICAL TRIAL: NCT02473848
Title: A Multi-center, Open-label, Uncontrolled, Investigator-initiated Trial to Evaluate the Safety and Efficacy of Ingenol Mebutate Gel 0.05% in Kidney Transplant Recipients With Actinic Keratoses on the Trunk and Extremities
Brief Title: Ingenol Mebutate Gel 0.05% in Kidney Transplant Recipients With Actinic Keratoses
Acronym: IMOT001
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of enrolment
Sponsor: Günther Hofbauer (Other)
Responsible Party: Sponsor-Investigator, Günther Hofbauer, Senior staff physician, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEKZH2013-0525
Record Dates: First submitted 2015-06-10; First posted 2015-06-17 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ingenol mebutate 500 ucg (Experimental): active arm
  Interventions: Drug: ingenol mebutate 500 ucg

INTERVENTIONS:
Drug: ingenol mebutate 500 ucg — Ingenol mebutate gel, 0.05%, commercially supplied in a box of 2 single use, unit dose tubes for topical application for each 25cm2, four conjunctive 25cm2 areas (100cm2) will be treated. If the 100 cm2 area is not cleared at Day 57 (+/- 3 Days), a second treatment cycle will be initiated with commercially supplied drug in a box of 2 single use, unit dose tubes for topical application for each 25cm2 and four conjunctive 25cm2 areas (100cm2 ) will be treated. In total for the first cycle, 4 commercially supplied boxes (8 unit dose tubes) will be used, and for the second cycle an additional 4 commercially supplied boxes (8 unit dose tubes) will be used (in total 8 boxes, 16 unit dose tubes per patient).
  Other Names: Picato 500 ucg

SUMMARY:
The substance ingenol mebutate (IM) is registered in Switzerland and many countries worldwide for the treatment of actinic keratosis (AK). There is no data on the use of IM in organ transplant recipients, a population highly affected by AK and skin cancer at large. The investigators want to study the use of IM against AK in this high-risk group of patients and assess its safety. The investigators are hoping to prove that IM is safe to use in AK of organ transplant recipients, allowing its use in the clinical routine treatement of AK also in this subset of patients with AK.

DETAILED DESCRIPTION:
Ingenol mebutate gel, 0.05%, commercially supplied in a box of 2 single use, unit dose tubes for topical application for each 25cm2, four conjunctive 25cm2 areas (100cm2) will be treated. If the 100 cm2 area is not cleared at Day 57 (+/- 3 Days), a second treatment cycle will be initiated with commercially supplied drug in a box of 2 single use, unit dose tubes for topical application for each 25cm2 and four conjunctive 25cm2 areas (100cm2 ) will be treated. In total for the first cycle, 4 commercially supplied boxes (8 unit dose tubes) will be used, and for the second cycle an additional 4 commercially supplied boxes (8 unit dose tubes) will be used (in total 8 boxes, 16 unit dose tubes per patient).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects 18 years of age or older
* Female subjects 18 years of age or older of non-child bearing potential defined by a serum follicle stimulating hormone (FSH) level ≥ 25.8 mIU/ml or by a confirmed clinical history of sterility (e.g. hysterectomy)
* Renal transplantation performed two years or more before inclusion
* Stable renal transplant function as determined by physician
* Actinic keratosis, one or multiple, of the trunk and/or extremities, non-hypertrophic non-hyperkeratotic based on clinical judgment within an area of 100 cm2 total (several areas adding up to 100 cm2 permissible)
* Signed Informed Consent after oral and written explanation of the study protocol

Exclusion Criteria:

* contraindications on ethical grounds such as inability to give informed consent
* women of child-bearing potential, women who are pregnant or breast feeding
* other clinically significant concomitant disease (e.g. hepatic dysfunction, cardiovascular disease, etc) at the investigator's discretion
* known or suspected non-compliance, drug or alcohol abuse
* enrolment into a clinical trial within last 4 weeks
* prior treatment with ingenol mebutate gel
* prior local/topical treatments in the treatment area within 2 weeks of trial entry:

  * Dermabrasion, chemical peeling, laser treatment, cryotherapy or surgery
  * Imiquimod, diclofenac, 5-Fluorouracil (5-FU), topical corticosteroids, topical retinoids, treatment with ultraviolet B (UVB) or photodynamic treatment (PDT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety (Change in creatinine from baseline) | 24 weeks
  Change in creatinine from baseline

SECONDARY OUTCOMES:
Efficacy (Reduction in actinic keratosis lesion count) | 24 weeks
  Reduction in actinic keratosis lesion count

CONTACTS AND LOCATIONS:
Overall Officials: Günther FL Hofbauer, MD, Principal Investigator — Dermatology Department University Hospital
Locations (1):
- Dermatology Department University Hospital Zürich, Zurich, Switzerland